CLINICAL TRIAL: NCT01068405
Title: Erosive Osteoarthritis of the Hands: Treatment by Methotrexate Versus Placebo - Assessment of Structural and Clinical Action of Magnetic Resonance Imaging
Brief Title: Erosive Osteoarthritis of the Hands: Treatment by Methotrexate Versus Placebo
Acronym: ADEM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-API-07
Record Dates: First submitted 2010-01-12; First posted 2010-02-15 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Polyarthritis
MeSH Terms: conditions — Arthritis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (Experimental): Patients with digital arthritis receiving methotrexate treatment at 10mg/week during 12 months
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Patients with digital arthritis receiving placebo at 10mg/week during 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate: 10mg/week administered in one time, the same day each week (every monday for example)during 12 months
  Arms: Methotrexate
Drug: Placebo — Placebo:10mg/week administered in one time, the same day each week (every monday for example)during 12 months
  Arms: Placebo

SUMMARY:
Interest of methotrexate in inflammatory rheumatisms was demonstrated since several years.

At present time,there is no effective treatment against digital arthritis. The investigators purpose to measure the efficacy of methotrexate on digital arthritis.

In this aim, two groups were compared. The first group receive 10mg/week of methotrexate administered in one shot (every Monday for example)during 12 months. The second group receive 10mg/week of placebo according to the same procedure

ELIGIBILITY:
Inclusion Criteria:

* hand arthritis
* pain over 40/100
* stable treatment since 4 weeks at least with non-steroid analgesic
* between 45 et 85 years

Exclusion Criteria:

* pregnancy or breast feeding women
* hyaluronic acid injection within the past 6 months
* cortisonic derivated injection within the past 3 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
pain assessed with EVA | at screening visit, inclusion visit, first month, and every month during one year

SECONDARY OUTCOMES:
Quality of life survey : SF-36 | at inclusion visit, first month, and every month during one year

CONTACTS AND LOCATIONS:
Overall Officials: Christian H ROUX, PhD, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Rheumatology Department, Nice, France

REFERENCES:
- [Derived] Ferrero S, Wittoek R, Allado E, Cruzel C, Fontas E, Breuil V, Ziegler L, Kremer J, Loeuille D, Roux CH. Methotrexate treatment in hand osteoarthritis refractory to usual treatments: A randomised, double-blind, placebo-controlled trial. Semin Arthritis Rheum. 2021 Aug;51(4):831-838. doi: 10.1016/j.semarthrit.2021.04.016. Epub 2021 May 6. PMID 34157578
- [Derived] Allado E, Wittoek R, Albuisson E, Ferrero S, Chenuel B, Chary-Valckenaere I, Roux C, Loeuille D. Topographical analysis of structural lesions between dominant and non-dominant hands in erosive osteoarthritis. Rheumatol Int. 2021 Mar;41(3):617-623. doi: 10.1007/s00296-020-04784-1. Epub 2021 Jan 27. PMID 33501510